CLINICAL TRIAL: NCT06614582
Title: Long-term Evaluation of Nasopharyngeal Airway in Hypotonia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Louise O'Brien, Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00239400
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Hypotonia, Muscle; Obstructive Sleep Apnea; Nasal Airway Obstruction
Keywords: Self-Supporting Nasopharyngeal Airway (ssNPA); Sleep study; Difficulty breathing; Obstructive Sleep Apnea; Cerebral Palsy; Down syndrome; Trisomy 21
MeSH Terms: conditions — Muscle Hypotonia; Sleep Apnea, Obstructive; Nasal Obstruction; Dyspnea; Cerebral Palsy; Down Syndrome

STUDY DESIGN:
Intervention Model Description: Single group intervention for participants who have completed NCT05527652 (Self-Supporting Nasopharyngeal Airway (ssNPA) Treating Upper Airway Obstruction in Hypotonia)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Self-Supporting Nasopharyngeal Airway (ssNPA) (Experimental): Participants will use the device up to 24 months.
  Interventions: Device: Self-Supporting Nasopharyngeal Airway (ssNPA)

INTERVENTIONS:
Device: Self-Supporting Nasopharyngeal Airway (ssNPA) — The ssNPA device is a flexible, medical-grade silicone, nasal tube that is self-inserted into the airway through one nostril and worn during the night. It can also be used during the day. The device works by supporting collapsed airway muscles and keeping the airway open.
  In addition to wearing the device, study team members will call monthly and collect certain data, and medical information and participants will be asked to have a sleep study at the 12-month visit.

SUMMARY:
This research is studying the long term use of a nasal airway device (self-supporting nasopharyngeal airway; "ssNPA") in children with hypotonic upper airway obstruction to learn about its effectiveness and tolerability as a treatment for obstructive sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* Children with Hypotonic Upper Airway Obstruction (HUAO) that took part in the original study (HUM00189669/NCT04846400 or HUM00220966/NCT05527652 trials)
* Willingness to continue device usage.
* Confirmed diagnosis of OSA (apnea/hypopnea index; AHI > 10 or AHI >5 with lowest oxygen level ≤75%)
* At least one symptom of OSA (such as frequent snoring, daytime sleepiness, or hyperactive/inattentive behaviors)
* Previous adenotonsillectomy (unless tonsillectomy not possible)
* Tonsil size 2+ or smaller

Exclusion Criteria:

* Participants that were non-compliant with the Self-Supporting Nasopharyngeal Airway (ssNPA) device during participation in the parent study listed above
* Any medical reason why ssNPA therapy may not be suitable
* Active COVID 19 infections Moderate/severe tracheobronchomalacia
* Need for anticoagulative therapy
* Bleeding disorder
* Restrictive thoracic disorders

Ages: 3 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Obstructive sleep apnea (OSA) severity measured by the apnea/hypopnea index (AHI) assessed by overnight polysomnography | Approximately 1 year
  Device efficacy will be measured by apnea/hypopnea index.
Long term device tolerability assessed by self-report from caregivers | 2 years
  This is a one question (likert scale 1-10) that participants' caregivers will complete at the final assessment (higher scores indicating better device tolerability).

SECONDARY OUTCOMES:
Long-term impact on sleep quality will be assessed by the mean score on the parent report of sleep quality | 1-2 years
  This will be a on a scale 1-10 (higher score is better).
Long-term impact on daytime sleepiness will be assessed by the mean score on the children's Epworth Sleepiness Scale (ESS) | 1-2 years
  The Epworth Sleepiness Scale is a self-administered form with eight items investigating sleep propensity in different real-life situations during the preceding months. Each item can receive 0-3 points, thus the final score ranges from 0 (best score) to 24 (worse score).
Long-term impact on quality of life will be assessed with the OSA-18 | 1-2 years
  This is an obstructive sleep apnea-specific quality of life tool for children and the Pediatric Quality of Life Inventory (PedsQL), a standard health-related quality of life instrument. Scores range from 0-126 with higher scores indicting worse impact. There are several dimensions of the PedsQL: Physical Functioning, Emotional Functioning, Social Functioning and School Functioning. Each domain will be scored on a scale of 0 (never have problems) to 4 (almost always have problems) and transformed on a scale of 0-100 by reverse scoring (0=100, 1=75, 2=50, 3=25, 4=0). Psychosocial Health Summary Score is the sum of the items over the number of items answered in the Emotional, Social, and School Functioning scales. Physical Health Summary Score is the Physical Functioning Scale Score. The total quality of life score is the sum of all the items over the number of items answered on all scales.
Family Impact Questionnaire (FIQ) | 1-2 years
  This tool measures parent's perceptions of the child's negative impact on the family. The FIQ is a 50-item, four-point Likert scale ranging from 0 (not at all) to 3 (very much) that asks about the impact the child has had on the family (e.g., social life, finances, marriage, and siblings) compared to the impact other children his/her age have on their families. Higher score is more significant impact.

CONTACTS AND LOCATIONS:
Overall Officials: Louise M O'Brien, PhD, MS, Principal Investigator — University Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Small number of complex children that could be identified by sharing Individual participant data (IPD).

REFERENCES:
- [Background] Powell AR, Srinivasan S, Helman JL, Li AD, O'Brien LM, Shih A, Plott JS, Zopf DA. Novel treatment for hypotonic airway obstruction and severe obstructive sleep apnea using a nasopharyngeal airway device with 3D printing innovation. J Clin Sleep Med. 2022 Oct 1;18(10):2497-2502. doi: 10.5664/jcsm.10202. PMID 35866230